CLINICAL TRIAL: NCT04394897
Title: Total Intravenous Anesthesia With Remifentanil-propofol Admixture Using Single-infusion Technique
Brief Title: Total Intravenous Anesthesia With Remifentanil-propofol Admixture
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: Bezmialem VU
Record Dates: First submitted 2020-04-09; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Total Intravenous Anesthesia; Propofol; Remifentanil; Bispectral Index Monitoring

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TIVA: TIVA either with remifentanil and propofol infusions separately
- MIXTIVA 2/1000: MIXTIVA infusion that had remifentanil/propofol proportion 2/1000
  Interventions: Combination Product: Remifentanil-Propofol admixture
- MIXTIVA 3/1000: MIXTIVA infusion that had remifentanil/propofol proportion 3/1000
  Interventions: Combination Product: Remifentanil-Propofol admixture

INTERVENTIONS:
Combination Product: Remifentanil-Propofol admixture
  Groups: MIXTIVA 2/1000; MIXTIVA 3/1000

SUMMARY:
Background: Application of total intravenous anesthesia (TIVA) may be considered as unpractical when compared with inhalational anesthesia. Although it is mostly not recommended, mixing intravenous agents seems to be popular in clinical practice. The aim of the study was to investigate the possible clinical drawbacks of using remifentanil-propofol admixture (MIXTIVA) for TIVA.

DETAILED DESCRIPTION:
ASA I-II adult patients scheduled for elective thyroidectomy were randomly allocated into 3 groups (n= 32 for each) to have TIVA either with remifentanil and propofol infusions separately (control group, Group I) or with MIXTIVA infusion that had remifentanil/propofol proportion 2/1000 or 3/1000 (remifentanil concentration 20 µg/ml or 30 µg/ml in propofol 1%, Group II or Group III respectively).

This technique may be considered as a practical implementation for busy ambulatory surgery centers performing general anesthesia, but delayed recovery may be predicted with longer duration of surgery and anesthesia.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiologists (ASA) physical status I patients American Society of Anesthesiologists (ASA) physical status II patients

Exclusion Criteria:

American Society of Anesthesiologists (ASA) physical status III patients or above patients A body mass index >35 kg/m2 Pregnant patients Breast-feeding Menstruating women Patients who were not euthyroid Uncontrolled hypertension Hepatic, renal or cardiac insufficiency Alcohol, opioid or drug abuse Allergy or contraindication to any of the study drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA I-II adult patients scheduled for elective thyroidectomy were randomly allocated into 3 groups (n= 32 for each)
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2013-03-12 (Actual); Primary Completion 2014-04-12 (Actual); Study Completion 2014-04-12 (Actual)

PRIMARY OUTCOMES:
Heart Rate Changes | During the application of TIVA
  Bradycardia: heart rate <45 beat per / min
Blood Pressure Changes | During the application of TIVA
  Hypotension (MAP <60 mmHg), Hypertension( systolic arterial pressure >150 mmHg)
Bispectral Index (BIS) Changes | During the application of TIVA
  BIS levels >60

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson BJ, Bagshaw O. Practicalities of Total Intravenous Anesthesia and Target-controlled Infusion in Children. Anesthesiology. 2019 Jul;131(1):164-185. doi: 10.1097/ALN.0000000000002657. PMID 30920966
- [Background] Errando CL, Sigl JC, Robles M, Calabuig E, Garcia J, Arocas F, Higueras R, Del Rosario E, Lopez D, Peiro CM, Soriano JL, Chaves S, Gil F, Garcia-Aguado R. Awareness with recall during general anaesthesia: a prospective observational evaluation of 4001 patients. Br J Anaesth. 2008 Aug;101(2):178-85. doi: 10.1093/bja/aen144. Epub 2008 May 30. PMID 18515816
- [Background] Roberts FL, Dixon J, Lewis GT, Tackley RM, Prys-Roberts C. Induction and maintenance of propofol anaesthesia. A manual infusion scheme. Anaesthesia. 1988 Mar;43 Suppl:14-7. doi: 10.1111/j.1365-2044.1988.tb09061.x. PMID 3259089
- [Background] Lamperti M. Adult procedural sedation: an update. Curr Opin Anaesthesiol. 2015 Dec;28(6):662-7. doi: 10.1097/ACO.0000000000000244. PMID 26356290
- [Background] Weatherall A, Venclovas R. Experience with a propofol-ketamine mixture for sedation during pediatric orthopedic surgery. Paediatr Anaesth. 2010 Nov;20(11):1009-16. doi: 10.1111/j.1460-9592.2010.03420.x. PMID 20964766
- [Derived] Bakan M, Umutoglu T, Topuz U, Guler EY, Uysal H, Ozturk E. Prospective evaluation of remifentanil-propofol mixture for total intravenous anesthesia: A randomized controlled study. Exp Ther Med. 2021 Nov;22(5):1198. doi: 10.3892/etm.2021.10632. Epub 2021 Aug 23. PMID 34584543